CLINICAL TRIAL: NCT01441388
Title: A Phase 1B, Open-Label, Dose Escalation Study To Evaluate Safety, Pharmacokinetics And Pharmacodynamics Of Crizotinib (PF-02341066) Plus VEGF Inhibitor Combinations In Patients With Advanced Solid Tumors.
Brief Title: A Study Of Crizotinib Plus VEGF Inhibitor Combinations In Patients With Advanced Solid Tumors.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business/Operational issues
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8081030
Record Dates: First submitted 2011-09-23; First posted 2011-09-27 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Carcinoma, Renal Cell; Glioblastoma; Carcinoma, Hepatocellular
Keywords: Phase 1b; crizotinib; sunitinib; axitinib; sorafenib; bevacizumab; cMET inhibitor; VEGF inhibitor; crizotinib combination
MeSH Terms: conditions — Carcinoma, Renal Cell; Glioblastoma; Carcinoma, Hepatocellular | interventions — Crizotinib; Axitinib; Sunitinib; Bevacizumab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose Escalation (Experimental): Histological or cytological diagnosis of advanced/metastatic solid tumor that is resistant to standard therapy or for which no standard therapy is available.
  Interventions: Drug: Crizotinib plus VEGF inhibitor combinations
- Expansion Population 1 (Experimental): Patients with histologically confirmed metastatic renal cell cancer with no prior systemic therapy directed at the malignant tumor.
  Interventions: Drug: Crizotinib plus axitinib; Drug: Crizotinib plus sunitinib
- Expansion Population 2 (Experimental): Patients with histologically confirmed metastatic renal cell cancer whose prior systemic therapy directed at the malignant tumor was single agent VEGF inhibitor and who now have acquired resistance to this treatment.
  Interventions: Drug: Crizotinib plus axitinib; Drug: Crizotinib plus sunitinib
- Expansion Population 3 (Experimental): Patients with histologically confirmed glioblastoma whose disease has failed on previous therapy, and which must have included treatment with external beam radiation and temozolomide chemotherapy, and who now have radiographically recurrent or progressive disease.
  Interventions: Drug: Crizotinib plus bevacizumab
- Expansion Population 4 (Experimental): Patients with histologically confirmed advanced-stage (unresectable or metastatic) hepatocellular carcinoma who have not received previous systemic therapy directed at the malignant tumor will be eligible to receive crizotinib plus sorafenib, should this combination be tested.
  Interventions: Drug: Crizotinib plus sorafenib

INTERVENTIONS:
Drug: Crizotinib plus VEGF inhibitor combinations — Three combinations will be prioritized, namely crizotinib plus axitinib, crizotinib plus sunitinib and crizotinib plus bevacizumab, with a fourth combination, crizotinib plus sorafenib to be tested only if crizotinib does not combine with either axitinib and/or sunitinib. All study drugs are tablets or capsules except for bevacizumab which is parenteral (intravenous). Dosage, frequency and duration to be determined.
  Arms: Dose Escalation
Drug: Crizotinib plus axitinib — Study drugs are tablets or capsules; dosage, frequency and duration to be determined.
  Arms: Expansion Population 1
Drug: Crizotinib plus sunitinib — Study drugs are tablets or capsules; dosage, frequency and duration to be determined.
  Arms: Expansion Population 1
Drug: Crizotinib plus axitinib — Study drugs are tablets or capsules; dosage, frequency and duration to be determined.
  Arms: Expansion Population 2
Drug: Crizotinib plus sunitinib — Study drugs are tablets or capsules; dosage, frequency and duration to be determined.
  Arms: Expansion Population 2
Drug: Crizotinib plus bevacizumab — Study drugs are tablets or capsules except for bevacizumab which is parenteral (intravenous). Dosage, frequency and duration to be determined.
  Arms: Expansion Population 3
Drug: Crizotinib plus sorafenib — Study drugs are tablets or capsules; dosage, frequency and duration to be determined.
  Arms: Expansion Population 4

SUMMARY:
Despite the success of anti-angiogenic therapy in multiple treatment settings, a fraction of patients are refractory to vascular endothelial growth factor (VEGF) inhibitor treatment while the majority of patients will eventually develop evasive resistance and exhibit disease progression while on therapy. It is proposed that mesenchymal-epithelial transition factor (c-MET) and its ligand hepatocyte growth factor (HGF or scatter factor) contribute significantly to VEGF inhibitor resistance such that combining a c-MET inhibitor with a VEGF inhibitor will provide additional clinical activity compared to VEGF inhibitor alone. This hypothesis will be tested using the cMET/ALK inhibitor, crizotinib, in combination with individual VEGF inhibitors. Three combinations will be prioritized, namely crizotinib plus axitinib, crizotinib plus sunitinib and crizotinib plus bevacizumab, with a fourth combination, crizotinib plus sorafenib to be tested only if crizotinib does not combine with either axitinib and/or sunitinib.

ELIGIBILITY:
Inclusion Criteria:

* Dose Escalation Population: Histological or cytological diagnosis of advanced/metastatic solid tumor that is resistant to standard therapy or for which no standard therapy is available. Lesions may be measurable or non measurable.
* Expansion Population 1: Patients with histologically confirmed metastatic renal cell cancer with no prior systemic therapy directed at the malignant tumor.
* Expansion Population 2: Patients with histologically confirmed metastatic renal cell cancer whose prior systemic therapy directed at the malignant tumor was single agent VEGF inhibitor and who now have acquired resistance to this treatment. Resistance is defined as progression following an initial response (complete or partial), or stable disease for at least 6 months on single agent VEGF inhibitor.
* Expansion Population 3: Patients with histologically confirmed glioblastoma whose disease has failed on previous therapy, and which must have included treatment with external beam radiation and temozolomide chemotherapy, and who now have radiographically recurrent or progressive disease.
* Expansion Population 4: Patients with histologically confirmed advanced-stage (unresectable or metastatic) hepatocellular carcinoma who have not received previous systemic therapy directed at the malignant tumor will be eligible to receive crizotinib plus sorafenib, should this combination be tested. Eligibility criteria also include normal hepatic function or Child-Pugh hepatic function class A.

Exclusion Criteria:

* Patients with hemorrhagic brain metastases or with known symptomatic brain metastases requiring steroids.
* Major surgery within 4 weeks of starting study treatment.
* Radiation therapy within 2 weeks of starting study treatment.
* Hypertension that cannot be controlled with medications (>150/90 mmHg despite optimal medical therapy).
* For glioblastoma patients: Prior treatment of glioblastoma with Gliadel wafers, stereotactic radiation, or brachytherapy unless there is pathological or definitive radiological evidence (PET scan or perfusion MRI) of recurrent tumor or unless there is new enhancement outside of the radiation field. History of Grade 2 or greater acute intracranial hemorrhage. Radiation therapy (RT) for glioblastoma within 3 months unless there is either: a) histopathologic confirmation of recurrent tumor, or b) new enhancement on MRI outside of the RT treatment field.Concomitant treatment with therapeutic doses of anticoagulants (low dose warfarin (Coumadin) up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs). | 12 months

SECONDARY OUTCOMES:
Duration of Response (DR) | 24 months
Progression free survival (PFS) | 24 months
Area under the plasma concentration versus time curve (AUC) of crizotinib and each VEGF inhibitor | 24 months
Best overall response, as assessed using the Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1 or , in the case of GBM (glioblastoma multiforme , RANO (Response Assessment in Neuro-Oncology) criteria. | 24 months
Overall survival (OS) up to 12 months | 24 months
Pre- and post-dose levels of soluble peripheral blood biomarkers. | 24 months
Tumor tissue biomarkers. | 18 months
6-month progression free survival proportion (PFS6) for glioblastoma patients | 24 months
Peak plasma concentration (Cmax) of crizotinib and each VEGF inhibitor | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081030&StudyName=A%20Study%20Of%20Crizotinib%20Plus%20VEGF%20Inhibitor%20Combinations%20In%20Patients%20With%20Advanced%20Solid%20Tumors.